CLINICAL TRIAL: NCT01326598
Title: Effectiveness of V-Go™ for Patients With Diabetes in a Real-world Setting: A Long-term, Prospective, Observational Registry (SIMPLE)
Brief Title: Effectiveness of V-Go™ for Patients With Diabetes in a Real-world Setting
Acronym: SIMPLE
Status: Completed | Type: Observational
Sponsor: Valeritas, Inc. (Industry)
Collaborators: Integrated Medical Development (Industry)
Responsible Party: Sponsor
Other Study IDs: V4006
Record Dates: First submitted 2011-03-03; First posted 2011-03-31 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: V Go™; Type 2 Diabetes; Insulin; Oral Anti Hypoglycemic Drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- T2DM patients with A1C<7.0%
  Interventions: Device: V-Go™

INTERVENTIONS:
Device: V-Go™ — Use of Insulin Delivery Device, V-Go, and the effect on A1C for T2DM patients in five categories of baseline oral antidiabetes drug (OAD) use with or without insulin.

SUMMARY:
The aim of the present study is to observe glycemic control, dose requirements, hypoglycemia risk, other possible adverse effects and weight changes, as well as to compare these parameters to prior treatment when patients with type 2 diabetes are initiated and treated using V-Go during circumstances as close to normal clinical practice as possible.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed type 2 diabetes mellitus for at least 12 months.
2. Must be and have been in stable treatment for at least a month within each of the following diabetes medication regimens:

   * OADs only,
   * OADs in combination with either exenatide, pramlintide, liraglutide (collectively termed "incretin mimetics") without receiving insulin,
   * Once or twice daily injection of an intermediate or long acting insulin (insulin NPH, insulin detemir or insulin glargine) with or without OADs and/or an incretin.
   * One to three daily injections of premix insulin (human insulin 70/30, insulin lispro 75/25 or insulin aspart 70/30) with or without OADs and/or an incretin.
   * Any insulin therapy with three or more insulin injections a day with or without OADs (MDI).
3. Must be willing to self monitor glucose at least twice a day.
4. The patient must be willing and able in the opinion of the investigator to try V-Go as therapy.
5. Age between 21 and 80 years old, inclusive.
6. A1C greater than or equal to 7.0%.

Exclusion Criteria:

1. Acute infection with fever.
2. Serum creatinine > 3.0 mg/dl if not on metformin, or if on metformin for females creatinine > 1.4 mg/dl, for males creatinine > 1.5 mg/dl within the last 6 months.
3. Pregnancy, intention to become pregnant or failure to agree to use adequate contraceptive measures during the trial for females of current reproductive potential.Medically acceptable contraceptives include: (1) surgical sterilization (such as tubal ligation or hysterectomy), (2) approved hormonal contraceptives (pills, patches, implants, or injections), (3) barrier methods (condom, diaphragm) used with spermicide, or (4) intrauterine device (IUD). Contraceptive measures such as "Plan B™", for emergency use after unprotected sex, are not acceptable methods for routine use. A lifestyle of abstinence from sexual activity is an acceptable means of contraception. If currently abstinent, the subject must agree to use a double-barrier method as described above if they become sexually active during the study period.
4. Any medical history of malignant melanoma or breast cancer.
5. Medical history of any other cancers within the last five years except adequately treated basal cell carcinoma or cervical carcinoma in-situ.
6. History of alcohol or drug abuse within the last year.
7. Any medical condition that in the opinion of the investigator may preclude safe and successful completion of the trial.
8. Participation in other clinical trials involving receipt of investigational drug that cannot be disclosed within the last 30 days.
9. Unwillingness and/or inability to comply with study procedures.
10. Require regular adjustments or modifications to the basal rate during a 24-hour period, or if the amount of insulin used at meals require adjustments of less-than 2-Unit increments.
11. History of hypersensitivity or hyperreactivity to adhesives.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes Mellitus
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare change of average glycemic control as measured by A1C from baseline to the end of V-Go use for the whole cohort as well as each of the five categories of baseline treatment. | 12 month

SECONDARY OUTCOMES:
Glycemic control is measured by the HbA1C from the beginning of the study to the end. | 12 month
  To describe change of average glycemic control as measured by A1C from baseline to the particular time point of analysis irrespective of treatment, and to describe this change for subjects who are still treated with the V-Go and those who have switched to other therapies.
To describe the incidence of hypoglycemia in participants as measured by blood glucose of <70 mg/dl. | 12 month
  Occurrence of hypoglycemia confirmed with self monitored plasma referenced glucose measurement <70 mg/dl.
Number of Participants with adverse events. | 12 month
How well the participants follow their doctors prescriptions for diabetes care. | 12 month
  To describe frequency of self monitoring plasma glucose with V-Go therapy
To describe insulin dose requirements from the beginning to the end of the study , and concomitant drugs to lower blood glucose. | 12 month
  Some of the insulin dose requirement that will described are: starting dose, dose titration, basal rate selection, dose conversion from previous therapy.
To describe changes in participants' weight from the beginning to the end of the study. | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Bohannon, MD, Principal Investigator — Nancy J. Bohannon Med. Corp; David Huffman, MD, Principal Investigator — University Diabetes & Endocrine Consultants; George Grunberger, MD, Principal Investigator — Grunberger Diabetes Institute; Kenneth Hershon, MD, Principal Investigator — North Shore Diabetes & Endocrine Assoc.; Chip Reed, MD, Principal Investigator — Endocrine Research Solutions, Inc.; Cheryl Rosenfeld, DO, Principal Investigator — North Jersey Endocrine Consultants, LLCAND; Alan B. Schorr, DO, Principal Investigator — Alan B. Schorr, DO FACE; Mark Warren, MD, Principal Investigator — Physicians East, PA; Richard A. Guthrie, MD, Principal Investigator — MidAmerica Diabetes Associates; Lenita Hanson, MD, Principal Investigator — MEDSOL Clinical Research Center; Philip A. Levin, MD, Principal Investigator — MODEL Clinical Research; Michael Shanik, MD, Principal Investigator — Endocrine Associates of Long Island, PC; Kathryn Jean Lucas, MD, Principal Investigator — Diabetes & Endocrinology Consultants; Mary Katherine Lawrence, MD, Principal Investigator — Down East Medical Associates; Sherry Sussman, MD, Principal Investigator — Middle Country Endocrinology, P.C.; Robert Bernstein, MD, Principal Investigator — Regional Endocrinology Associates, PC; Albert Johary, MD, Principal Investigator — Albert Johary M.D., P.C.; Jeffrey Rothman, MD, Principal Investigator — University Physicians Group; Robert Savino, DO, Principal Investigator — Western Connecticut Health Network, Inc.; Sarah Khan, MD, Principal Investigator — Parsippany Endocrine, LLC; Jonathan Wilson, DO, Principal Investigator — PMG Research of Winston-Salem; Stephanie Powell, MD, Principal Investigator — PMG Research of Bristol; Rickey Manning, MD, Principal Investigator — PMG Research of Knoxville; Georges M. Argoud, MD, Principal Investigator — San Diego Coastal Endocrinology Group
Locations (25):
- United States (25):
  - San Diego Coastal Endocrinology Group, Chula Vista, California
  - Nancy J. Bohannon Med. Corp, San Francisco, California
  - Western Connecticut Health Network, Inc., Danbury, Connecticut
  - MEDSOL Clinical Research Center, Port Charlotte, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Albert Johary M.D., P.C., Dunwoody, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - MidAmerica Diabetes Associates, Wichita, Kansas
  - MODEL Clinical Research, Baltimore, Maryland
  - Grunberger Diabetes Institute, Bloomfield Hills, Michigan
  - North Jersey Endocrine Consultants, LLCAND, Denville, New Jersey
  - Parsippany Endocrine, LLC, Parsippany, New Jersey
  - Regional Endocrinology Associates, PC, Santa Fe, New Mexico
  - North Shore Diabetes & Endocrine Assoc., New Hyde Park, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - Middle Country Endocrinology, P.C., Smithtown, New York
  - University Physicians Group, Staten Island, New York
  - Physicians East, PA, Greenville, North Carolina
  - Diabetes & Endocrinology Consultants, Morehead City, North Carolina
  - Down East Medical Associates, Morehead City, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Alan B. Schorr, DO FACE, Langhorne, Pennsylvania
  - PMG Research of Bristol, Bristol, Tennessee
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee

REFERENCES:
- [Derived] Grunberger G, Rosenfeld CR, Bode BW, Abbott SD, Nikkel C, Shi L, Strange P. Effectiveness of V-Go(R) for Patients with Type 2 Diabetes in a Real-World Setting: A Prospective Observational Study. Drugs Real World Outcomes. 2020 Mar;7(1):31-40. doi: 10.1007/s40801-019-00173-8. PMID 31833010
- See also: V-Go™ — http://www.valeritas.com